CLINICAL TRIAL: NCT03921307
Title: Clinical Performance of Monolithic Lithium-disilicate Glass-Ceramic CAD/CAM Crowns
Brief Title: Clinical Performance of Ceramic CAD/CAM Crowns
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Ahmed Alamri, Assistant Professor, University of Toronto
Other Study IDs: 33291
Record Dates: First submitted 2019-04-07; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Tooth Crown Fracture; Dental Caries
Keywords: Computer-Aided Design; dental crowns; survival
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to evaluate the clinical performance of laboratory and chairside fabricated monolithic anterior and posterior LDGC CAD/CAM crowns performed by predoctoral students at the University of Toronto and the effect of different patient and provider-related factors on their longevity and to compare them to the metal-ceramic (MC) crowns. A sample of LDGC CAD/CAM crowns (IPS e.max, Ivoclar Vivadent) provided by predoctoral students was evaluated. Crown preparations were made according to the specific criteria and were milled in-house using the CEREC bluecam and Omnicam systems. Crowns were cemented with Rely-X Unicem (3M/ESPE) and Calibra Universal (Dentsply Sirona) resin cements. Clinical assessment of the crowns and supporting periodontal structures was performed following the modified California Dental Association (CDA) criteria. Intra-oral photographs, periapical and bitewing radiographs were taken for further assessment by two evaluators. Two-hundred and fifty-one patients with 275 crowns were examined with a follow-up period of up to 6 years.

DETAILED DESCRIPTION:
The clinical success of the monolithic Lithium-disilicate Glass-ceramic (LDGC) crowns manufactured with computer-aided design (CAD) / computer-aided manufacturing (CAM) technology provided by predoctoral students was not investigated. Thus, the purpose of this study was to evaluate the clinical performance of laboratory and chairside fabricated monolithic anterior and posterior LDGC CAD/CAM crowns performed by predoctoral students at the University of Toronto and the effect of different patient and provider-related factors on their longevity and to compare them to the metal-ceramic (MC) crowns. A sample of LDGC CAD/CAM crowns (IPS e.max, Ivoclar Vivadent) provided by predoctoral students was evaluated. Crown preparations were made according to the specific criteria and were milled in-house using the CEREC bluecam and Omnicam systems. Crowns were cemented with Rely-X Unicem (3M/ESPE) and Calibra Universal (Dentsply Sirona) resin cements. Clinical assessment of the crowns and supporting periodontal structures was performed following the modified California Dental Association (CDA) criteria. Intra-oral photographs, periapical and bitewing radiographs were taken for further assessment by two evaluators. Two-hundred and fifty-one patients with 275 crowns were examined with a follow-up period of up to 6 years. Part 1 evaluated the performance of laboratory-fabricated LDGC CAD/CAM crowns. Part 2 evaluated the performance of chairside LDGC CAD/CAM crowns. Forty crowns were evaluated. Part 3 evaluated the performance of LDGC CAD/CAM and MC crowns using split-mouth design. A total of 25 patients and 50 crowns (25 crowns for each group) were examined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy periodontal tissue Adequate root canal treatment

Exclusion Criteria:

* Parafunctional habits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who received dental treatment at the Faculty of Dentistry, University of Toronto.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Survival percentage | 6 years
  Kaplan Meier analysis of survival of the crowns
Clinical performance of crowns via modified California Dental Association (CDA) criteria | 6 years
  Biological complications: pulpal involvement, recurrent caries, tooth fracture. Technical complications: marginal integrity (slight marginal discrepancy, open margins, marginal overhang, under-contoured margins), loss of retention, crown fracture, chipping/crack lines, open proximal contact. Esthetic complications: surface texture/smoothness, color match/mismatch, marginal discoloration, over or under-contoured.

SECONDARY OUTCOMES:
Patient satisfaction with esthetic and function of crowns | 6 years
  Using Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Alamri, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altamimi AM, Tripodakis AP, Eliades G, Hirayama H. Comparison of fracture resistance and fracture characterization of bilayered zirconia/fluorapatite and monolithic lithium disilicate all ceramic crowns. Int J Esthet Dent. 2014 Spring;9(1):98-110. PMID 24757702
- [Background] Belli R, Petschelt A, Hofner B, Hajto J, Scherrer SS, Lohbauer U. Fracture Rates and Lifetime Estimations of CAD/CAM All-ceramic Restorations. J Dent Res. 2016 Jan;95(1):67-73. doi: 10.1177/0022034515608187. Epub 2015 Oct 1. PMID 26428908
- [Background] Cortellini D, Canale A. Bonding lithium disilicate ceramic to feather-edge tooth preparations: a minimally invasive treatment concept. J Adhes Dent. 2012 Feb;14(1):7-10. doi: 10.3290/j.jad.a22708. PMID 22282749
- [Background] Fasbinder DJ, Dennison JB, Heys D, Neiva G. A clinical evaluation of chairside lithium disilicate CAD/CAM crowns: a two-year report. J Am Dent Assoc. 2010 Jun;141 Suppl 2:10S-4S. doi: 10.14219/jada.archive.2010.0355. PMID 20516109
- [Background] Rauch A, Reich S, Dalchau L, Schierz O. Clinical survival of chair-side generated monolithic lithium disilicate crowns:10-year results. Clin Oral Investig. 2018 May;22(4):1763-1769. doi: 10.1007/s00784-017-2271-3. Epub 2017 Nov 4. PMID 29103104
- [Background] Reich S, Fischer S, Sobotta B, Klapper HU, Gozdowski S. A preliminary study on the short-term efficacy of chairside computer-aided design/computer-assisted manufacturing- generated posterior lithium disilicate crowns. Int J Prosthodont. 2010 May-Jun;23(3):214-6. PMID 20552085
- [Background] Seydler B, Schmitter M. Clinical performance of two different CAD/CAM-fabricated ceramic crowns: 2-Year results. J Prosthet Dent. 2015 Aug;114(2):212-6. doi: 10.1016/j.prosdent.2015.02.016. Epub 2015 Apr 30. PMID 25935085